CLINICAL TRIAL: NCT05454722
Title: A Study to Evaluate the Performance of Adex Gel in the Treatment of Atopic Eczema Using SCORAD and Quality of Life Assessments.
Brief Title: A Study to Evaluate Adex Gel in the Treatment of Atopic Eczema.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dermal Laboratories Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DENI-06
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Atopic Eczema
Keywords: SCORAD; CDLQI; QoL
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adex Gel (Experimental): Dry Skin Emollient with Nicotinamide
  Interventions: Device: ADEX Gel

INTERVENTIONS:
Device: ADEX Gel — Emollient Gel with added anti-inflammatory

SUMMARY:
This is a prospective, open label, uncontrolled study which will be performed in multiple Primary Care (GP) centres, in approximately 60 children (aged 1 year to 15 years) who have moderate atopic eczema and who are not currently using oral or topical corticosteroids or immunomodulators and have not used them in the previous month.

Study patients will be asked to use Adex Gel three times daily, for 4 weeks instead of their usual emollient or as the first treatment for their condition, and without supplementary use of any oral or topical steroids or immunomodulators (unless this becomes unavoidable, see section 4.6.3). The Scoring Atopic Dermatitis (SCORAD) assessment will be performed by the investigator/ research nurse at baseline and then after 2 and 4 weeks of treatment. Patients or their parents/ guardians will be asked to complete the quality-of-life questionnaires (Children's Dermatology Life Quality Index (CDLQI) at baseline and after 4 weeks of treatment. Photographs, which will not include any identifiable features or details of the patient, of one eczema affected area will also be taken at baseline and again 4 weeks after treatment.

DETAILED DESCRIPTION:
Patients will be recruited by the General Practitioner (GP) surgeries using their databases to identify patients who are currently atopic eczema sufferers and are using mainly emollients (other than Adex Gel) to manage their condition. Patients or their parents/guardians will be contacted by the surgery to see if they would like to participate in this study and to establish whether they are currently or have been using oral or topical corticosteroids or other immunomodulators in the previous 1 month. Advertisements in the surgery may also be used as these may encourage new eczema sufferers to ask the doctor if they could participate in this study. As new eczema patients they would not currently be using steroids for their condition so would be deemed eligible for screening.

Patients and their parents/legal guardians will attend the screening and enrolment visit where parents/legal guardians will be asked to sign an informed consent form, and where appropriate the participant will sign an assent form, confirming their agreement to take part in the study. A number of questions will be asked about medical history and current medications as well as eligibility criteria. No washout period will be implemented.

Those who are considered eligible to participate in accordance with the inclusion and exclusion criteria given in section 4.6, will then undergo their baseline assessments where the Investigator/ research nurse will perform the SCORAD assessments and record these in the patient's paper Case Report Form (CRF). The patient or their parent/ guardian will also complete a baseline quality of life questionnaire (CDLQI) and photographs will also be taken.

The patients will then be given sufficient supplies of Adex Gel (depending on the coverage of their eczema) to use over the 4 week use period (additional packs may be provided at visit 2, if necessary). They will be asked to use Adex Gel instead of their usual emollient (if already using one) and to try and refrain from using oral or topical corticosteroids, or immunomodulators for the duration of the study. If, in the opinion of the investigator, it becomes necessary for patients to use oral or topical corticosteroids or immunomodulators during the study, the Investigator/ research nurse will record this on their CRF, and the patient will be withdrawn from the study. Patients will be asked to record use of any other medication or topical products during the study in their Patient Diary.

After 2 weeks of treatment, patients will return to the GP surgery and will be asked about their compliance with the study requirements, changes in health and medications and any incidents will be recorded. They will again have their eczema assessed by the Investigator/ research nurse and the results recorded on the CRF.

After 4 weeks of treatment, patients will return to the surgery, where again they will be asked about compliance, changes in health and medications and any incidents will be recorded. They will also undergo their final Investigator/ research nurse assessment, have the area, which was selected at baseline, photographed, and complete the final quality-of-life questionnaire.

This visit will conclude their participation in the study unless follow-up of any incidents is required.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Aged between 1 year and 15 years.
* Patients with atopic eczema (personal or combined personal and familial atopy), of moderate severity in accordance with the NICE categorisation
* SCORAD assessment score of between 25 to 50.
* Minimum score of 6 on the CDLQI (QoL).
* Patients or their parents/ legal guardians must be able to read and understand the patient information sheet and sign the consent form.
* Patients normally managing their eczema by regular and ongoing use of leave-on emollient(s), or new atopic eczema sufferers, who have not been using oral or topical corticosteroids, Adex Gel or immunomodulators for the last month.
* Patients who are willing to use only Adex Gel for 4 weeks.
* Patients who are willing to continue to use their standard wash regime for the duration of the study. This will be documented at the initial visit.

Exclusion Criteria:

* Under 1 year of age or over 15 years and 11 months at screening.
* Are currently using or have used in the past month, any oral or topically applied corticosteroids, Adex Gel or immunomodulators for their atopic eczema.
* Have a known history of intolerance or skin sensitivity to any of the ingredients of Adex Gel (as identified on the patient information sheet and product labelling), or similar products.
* Have mild eczema.
* Have severe or potentially infected eczema.
* Participating in other ongoing studies or have participated in a study in the previous 30 days.
* Patients, or their parents/ legal guardians, who may have difficulties completing the quality-of-life questionnaire, which will be written in English only.
* Employees of the Sponsor or Investigators, or any immediate family member (partner, offspring, parents, siblings, or sibling's offspring) of such employees.
* Patients with any medical condition which, in the opinion of the Investigator, may adversely influence their participation in the study.

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
SCORAD | 4 weeks
  Change in SCORAD (SCORing Atopic Dermatitis, based on Area, Intensity and Subjective score. (Score of 0-103 with the higher the score the more severe the condition)) over 4 weeks.
QoL | 4 Weeks
  Change in CDLQI (Child Dermatology Quality of Life Index (a maximum score of 30 and a minimum score of 0. The higher the score, the more quality of life is effected)) over 4 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Cripps Health Centre, Nottingham, Nottinghamshire
  - Atherstone Surgery, Atherstone, Warwickshire

IPD SHARING:
Plan to Share IPD: No